CLINICAL TRIAL: NCT00395811
Title: Stem Cell Therapy to Improve Myocardial Function in Patients Undergoing Coronary Artery Bypass Grafting (CABG)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: China National Center for Cardiovascular Diseases, China National Center for Cardiovascular Diseases
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCCD200601
Record Dates: First submitted 2006-11-01; First posted 2006-11-03 (Estimated); Last update posted 2008-10-29 (Estimated); Status verified 2008-10

CONDITIONS: Coronary Disease; Myocardial Infarction
Keywords: Myocardial Infarction; stem cell therapy; Coronary Artery Bypass Grafting
MeSH Terms: conditions — Coronary Disease; Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Bone Marrow Stem Cell Therapy combined CABG — Bone Marrow Stem Cell inject into myocardium

SUMMARY:
The purpose of this study is to determine whether intracoronary transfer of autologous bone marrow cells can induce angiogenesis, subsequently improving regional myocardial perfusion, and finally resulting in improved systolic and diastolic left ventricular function in patients with myocardial infarction.

50 patients with stable left ventricle function will - with six months interval - receive two treatments with bone marrow transplantation intracoronary in vessels supplying dysfunctional myocardial territories and Coronary Artery Bypass Graft (CABG).

DETAILED DESCRIPTION:
This research study is being performed to find out more information about the safety and efficacy of autologous bone marrow stem cells transplantation. In patients with myocardial infarction, the heart muscle does not pump well. Over a period of years, this continues to get worse until the patient dies of heart failure. The researchers are trying to find out if the transplantation of these stem cell can make a change in the functioning of these areas of the heart muscle.

Patients between 18 and 70 years of age who received autologous bone marrow stem cell transplant at the Fuwai cardiovascular hospital may be eligible for this study. Candidates must have had their first transplant at least 3 years before entering the current study.

These patients receive autologous bone marrow cells transplantation intracoronary undergoing Coronary Artery Bypass Graft. The objective evaluations will be performed at baseline and during 6 months follow-up.

Heart function tests may include the following:

1. Electrocardiogram (EKG) evaluates the electrical activity of the heart. Electrodes placed on the chest transmit information from the heart to a machine.
2. Echocardiogram (Echo) is an ultrasound test that uses sound waves to create an image of the heart and examine the function of the heart chambers and valves.
3. Gated acquisition scan is a nuclear medicine test that uses a small amount of radioactive chemical injected into a vein. A special scanner creates an image of the heart for examining the beating motion of the muscle.
4. MRI evaluates function of the heart chambers the beating motion of the muscle.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with coronary disease undergoing CABG.
2. At least 3 months since last episode of myocardial infarction
3. Patients fulfilling either of the following criteria based on the extent of CAD by coronary angiography and LVEF by echocardiography.

   Reversible myocardial ischemia as revealed by SPECT. ejection fraction >=40% <=50%. Age >=18 years and <=70 Patients who can give informed consent themselves in writing.
4. Negative pregnancy test (in women with childbearing potential).

Exclusion Criteria:

Any one of the following exclusion criteria is sufficient to disqualify a patient from the study.

1. Sustained ventricular tachycardia in a 24-hour ECG.
2. Chronic atrial fibrillation.
3. Less than 3 months since last episode of cerebral infarction.
4. Patients with a malignant tumor*.
5. Patients with chronic rheumatoid arthritis.
6. Patients with a history of severe allergic reactions.
7. Patients with hematological disease (leukemia, myeloproliferative disease, or myelodysplastic syndromes).
8. Patients currently suffering from or having a history of interstitial pneumonitis.
9. Leukocytes less than 4,000/µL or exceeding 10,000/µL.
10. Platelets less than 100,000/µL.
11. Hemoglobin less than 10 g/dL.
12. AST (GOT) exceeding 100 IU/L or ALT (GPT) exceeding 100 IU/L.
13. Patients for whom it is impossible to perform both cardiac MRI
14. Pregnant or nursing patients, those who may be pregnant, or those who plan on becoming pregnant before the end of the study period.
15. Any other reason that the Clinical Supervisors or Clinical Researchers may have for considering a case unsuitable for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-01; Primary Completion 2009-04 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Changes in left ventricular ejection fraction from baseline to 6 months' follow-up | 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Hu shengshou, Study Director — National center for cardiovascular disease ,china
Locations (1):
- Fuwai cardiovascular disease hospital, Beijing, China

REFERENCES:
- [Derived] Hu S, Liu S, Zheng Z, Yuan X, Li L, Lu M, Shen R, Duan F, Zhang X, Li J, Liu X, Song Y, Wang W, Zhao S, He Z, Zhang H, Yang K, Feng W, Wang X. Isolated coronary artery bypass graft combined with bone marrow mononuclear cells delivered through a graft vessel for patients with previous myocardial infarction and chronic heart failure: a single-center, randomized, double-blind, placebo-controlled clinical trial. J Am Coll Cardiol. 2011 Jun 14;57(24):2409-15. doi: 10.1016/j.jacc.2011.01.037. PMID 21658561